CLINICAL TRIAL: NCT06433752
Title: REal World ExperieNce With BRIUMVI® (UblituximAB-xiiy) Treated Patients: A Longitudinal REgistry Study (ENABLE)
Brief Title: A Study Evaluating the Real World Experience of Participants Treated With BRIUMVI® (Ublituximab-xiiy) for Relapsing Multiple Sclerosis (RMS)
Acronym: ENABLE
Status: Recruiting | Type: Observational
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TG1101-RMS406
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BRIUMVI® (Ublituximab-xiiy): Participants will receive BRIUMVI® (Ublituximab-xiiy) intravenous (IV) infusion for the treatment of RMS.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The purpose of this study is to evaluate safety, effiectiveness, and to gain insight into the treatment experience of participants prescribed BRIUMVI® (ublituximab-xiiy) in the real-world setting

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed Multiple Sclerosis (MS) diagnosis.
2. Participants who have not received any BRIUMVI® (ublituximab-xiiy) infusion prior to study start. Participants who have been prescribed BRIUMVI® (ublituximab-xiiy) but have not yet received their first infusion on Day 1 of 150 milligrams (mg) can be included.

Exclusion Criteria:

1. Have received any live or live-attenuated vaccines (including for varicella-zoster virus or measles) within 4 weeks prior to first BRIUMVI® (ublituximab-xiiy) administration or any non-live vaccines within 2 weeks prior to first BRIUMVI® (ublituximab-xiiy) administration.
2. Any active infection (e.g., active Hepatitis B virus [HBV])
3. Concurrent participation in any interventional MS trials, or planned concurrent treatment with other Multiple Sclerosis Disease Modifying Therapy (MS DMT) during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants with RMS who are receiving BRIUMVI® (ublituximab-xiiy).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Annualized Relapse Rate (ARR) | Up to Week 96

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to Week 96
Number of Participants with Infusion Related Reaction (IRR) at Each Infusion | Up to Week 96

CONTACTS AND LOCATIONS:
Locations (74):
- United States (73):
  - TG Therapeutics Investigational Trial Site, Birmingham, Alabama
  - TG Therapeutics Investigational Trial Site, Mobile, Alabama
  - TG Therapeutics Investigational Trial Site, Gilbert, Arizona
  - TG Therapeutics Investigational Trial Site, Phoenix, Arizona
  - TG Therapeutics Investigational Trial Site, Scottsdale, Arizona
  - TG Therapeutics Investigational Trial Site, Newport Beach, California
  - TG Therapeutics Investigational Trial Site, Orange, California
  - TG Therapeutics Investigational Trial Site, West Hollywood, California
  - TG Therapeutics Investigational Trial Site, Aurora, Colorado
  - TG Therapeutics Investigational Trial Site, Basalt, Colorado
  - TG Therapeutics Investigational Trial Site, Colorado Springs, Colorado
  - TG Therapeutics Investigational Trial Site, Denver, Colorado
  - TG Therapeutics Investigational Trial Site, Fort Collins, Colorado
  - TG Therapeutics Investigational Trial Site, Grand Junction, Colorado
  - TG Therapeutics Investigational Trial Site, Farmington, Connecticut
  - TG Therapeutics Investigational Trial Site, Hartford, Connecticut
  - TG Therapeutics Investigational Trial Site, Wilmington, Delaware
  - TG Therapeutics Investigational Trial Site, Washington D.C., District of Columbia
  - TG Therapeutics Investigational Trial Site, Altamonte Springs, Florida
  - TG Therapeutics Investigational Trial Site, Boca Raton, Florida
  - TG Therapeutics Investigational Trial Site, Clearwater, Florida
  - TG Therapeutics Investigational Trial Site, Maitland, Florida
  - TG Therapeutics Investigational Trial Site, Miami, Florida
  - TG Therapeutics Investigational Trial Site, Naples, Florida
  - TG Therapeutics Investigational Trial Site, Weston, Florida
  - TG Therapeutics Investigational Trial Site, Atlanta, Georgia
  - TG Therapeutics Investigational Trial Site, Coeur d'Alene, Idaho
  - TG Therapeutics Investigational Trial Site, Chicago, Illinois
  - TG Therapeutics Investigational Trial Site, Evanston, Illinois
  - TG Therapeutics Investigational Trial Site, Urbana, Illinois
  - TG Therapeutics Investigational Trial Site, Lexington, Kentucky
  - TG Therapeutics Investigational Trial Site, Louisville, Kentucky
  - TG Therapeutics Investigational Trial Site, Baltimore, Maryland
  - TG Therapeutics Investigational Trial Site, Glen Burnie, Maryland
  - TG Therapeutics Investigational Trial Site, Boston, Massachusetts
  - TG Therapeutics Investigational Trial Site, Burlington, Massachusetts
  - TG Therapeutics Investigational Trial Site, Norfolk, Massachusetts
  - TG Therapeutics Investigational Trial Site, Ann Arbor, Michigan
  - TG Therapeutics Investigational Trial Site, Farmington, Michigan
  - TG Therapeutics Investigational Trial Site, Owosso, Michigan
  - TG Therapeutics Investigational Trial Site, Omaha, Nebraska
  - TG Therapeutics Investigational Trial Site, Las Vegas, Nevada
  - TG Therapeutics Investigational Trial Site, Freehold, New Jersey
  - TG Therapeutics Investigational Trial Site, Livingston, New Jersey
  - TG Therapeutics Investigational Trial Site, Neptune City, New Jersey
  - TG Therapeutics Investigational Trial Site, Teaneck, New Jersey
  - TG Therapeutics Investigational Trial Site, Amherst, New York
  - TG Therapeutics Investigational Trial Site, New York, New York
  - TG Therapeutics Investigational Trial Site, Charlotte, North Carolina
  - TG Therapeutics Investigational Trial Site, New Bern, North Carolina
  - TG Therapeutics Investigational Trial Site, Raleigh, North Carolina
  - TG Therapeutics Investigational Trial Site, Centerville, Ohio
  - TG Therapeutics Investigational Trial Site, Cincinnati, Ohio
  - TG Therapeutics Investigational Trial Site, Cleveland, Ohio
  - TG Therapeutics Investigational Trial Site, Columbus, Ohio
  - TG Therapeutics Investigational Trial Site, Toledo, Ohio
  - TG Therapeutics Investigational Trial Site, Portland, Oregon
  - TG Therapeutics Investigational Trial Site, Bethlehem, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Knoxville, Tennessee
  - TG Therapeutics Investigational Trial Site, Nashville, Tennessee
  - TG Therapeutics Investigational Trial Site, Austin, Texas
  - TG Therapeutics Investigational Trial Site, Dallas, Texas
  - TG Therapeutics Investigational Trial Site, Edinburg, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas
  - TG Therapeutics Investigational Trial Site, Charlottesville, Virginia
  - TG Therapeutics Investigational Trial Site, Norfolk, Virginia
  - TG Therapeutics Investigational Trial Site, Vienna, Virginia
  - TG Therapeutics Investigational Trial Site, Kirkland, Washington
  - TG Therapeutics Investigational Trial Site, Morgantown, West Virginia
  - TG Therapeutics Investigational Trial Site, Greenfield, Wisconsin
  - TG Therapeutics Investigational Trial Site, Milwaukee, Wisconsin
  - TG Therapeutics Investigational Trial Site, Neenah, Wisconsin
  - TG Therapeutics Investigational Trial Site, Waukesha, Wisconsin
- TG Therapeutics Investigational Trial Site, Guaynabo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No